CLINICAL TRIAL: NCT06538584
Title: Caffeine Facilitates the Recovery of Dexmedetomidine Sedation for MRI in Pediatric Patients: a Randomized, Double-blinded and Placebo-controlled Pilot Study
Brief Title: Dex +/- Caffeine Sedation in a Post-MRI Recovery in a Pediatric Population
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB24-0210
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Enhanced Recovery After Surgery in a Pediatric Population
Keywords: Dexmedetomidine sedation; Caffeine citrate stimulant; Pediatric surgical population
MeSH Terms: interventions — caffeine citrate; Sodium Citrate

STUDY DESIGN:
Intervention Model Description: A randomized model with 2 arms/interventions consisting of caffeine v. saline placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexmedetomidine +/- Caffeine Sedation (Experimental): Eligible subjects will be given 15 mg/kg caffeine citrate (equivalent to ~5 mg/ kg caffeine base) ~ 15 min after terminating Dex's infusion.
  Interventions: Drug: Caffeine citrate 15mg/kg
- Dexmedetomidine +/- Placebo Sedation (Placebo Comparator): Eligible subjects will be given 9 mg/ml saline placebo) ~ 15 min after terminating Dex's infusion.
  Interventions: Drug: 0.9% Sodium Citrate

INTERVENTIONS:
Drug: Caffeine citrate 15mg/kg — Subjects will be randomized prior to surgery into one of the two study arms. One arm will receive 15mg/kg Caffeine citrate 15 minutes post surgery.
  Arms: Dexmedetomidine +/- Caffeine Sedation
Drug: 0.9% Sodium Citrate — Subjects will be randomized prior to surgery into one of the two study arms. One arm will receive 0.9% Sodium Citrate/kg 15 minutes post surgery.
  Arms: Dexmedetomidine +/- Placebo Sedation

SUMMARY:
Dexmedetomidine (Dex), a selective α2-adrenergic receptor agonist, is the most used sedative for procedural sedation in children and in pediatric Intensive Care Unit (PICU) because it is associated with less respiratory depression and also less neurotoxicity; rather Dex appears neuroprotective. Unfortunately, Dex is associated with very long emergence times and may cause bradycardia and hypotension. However, using sedation dosing guidelines (by consensus among SPS members) 1-3 mcg/kg bolus and a 1-2 mcg/kg/hour infusion, hemodynamic compromise is less significant and rarely requires intervention in these patients. With this Dex sedation protocol, these pediatric patients usually take an average of 45 minutes (30-60 minutes) to wake and become alert and up to 2 hours to be discharged.

Without reversal agents, emergence times from Dex sedation are slow. The prolonged recovery after Dex sedation for non-surgical procedures negatively affects throughput, thus increasing the cost of care. Patient safety and satisfaction suffer as a result. The children wake feeling tired and sluggish. The children don't feel back to normal for an extended period of time, which is not surprising given that the half-life for Dex metabolism in 2-3 hours in humans. However, using sedation dosing guidelines (by consensus among SPS members) 1-3 mcg/kg bolus and a 1-2 mcg/kg/hour infusion, hemodynamic compromise is less significant and rarely requires intervention in these patients. In humans, it has been found that caffeine at 7.5 mg/kg (15 mg caffeine citrate equivalent to 7.5 mg caffeine base) sped emergence from isoflurane anesthesia with minimal hemodynamic effects in healthy human volunteers.

The goal of this clinical trial is to determine whether caffeine will facilitate the recovery of Dex sedation after a Magnetic Resonance Imaging (MRI) procedure by measuring the time from the end of Dex infusion to the time meeting the discharge criteria.

DETAILED DESCRIPTION:
SCREENING DAY (-1-3) - PRIOR TO APPOINTMENT Only a single visit will take place prior to the MRI scan procedure. This will be done one to three days prior to the sedation procedure, via chart screening or on the day of the sedation and MRI procedure if the advanced review is not possible.

Once potentially appropriate subjects have been identified from the OR schedule for the next day, the study team will contact the anesthesia provider (resident, CRNA, attending) who is scheduled to treat that patient and explain to him/her about the research project and ask them to use a Sedline Brain Function Monitor for the case.

* Sedation team calls patient family with reminder about appointment and NPO instructions.
* Research pharmacy notified about potential patients.

DAY 0 - APPOINTMENT DAY On the day of the Magnetic Resonance Imaging (MRI) procedure in the preoperative holding area.

* Study consent or/and assent obtained by study team in the pre-sedation area.
* Study team notifies research pharmacy to prepare/deliver study drug

PRE-SEDATION

* Patient arrives in sedation suite
* RN rooms patient, obtains vitals (height, weight, heart rate, respiratory rate, blood pressure, 3-lead electrocardiogram [EKG], and temperature), reviews allergies, and asks health-related questions
* Physician (MD) called to room to complete patient history, physical examination, and review/sign sedation consent
* Sedation physician reviews sedation plan with nurse
* The sedation physician will be delegated by the Principal Investigator (PI) and be Institutional Review Board (IRB)-approved on this study to provide the study drug
* Sedation physician enters H+P/orders while nurse starts the peripheral IV (PIV) and prepares sedation medication
* Sedation physician returns to bedside for induction In explaining the research project to anesthesia providers, the study team will stress the importance of keeping the patient's Sedline Density Spectral Array (DSA) between 8-15 or/and Patient State Index (PSI) reading between 25-50 throughout the course of the case in the subjects who are randomly selected in the monitoring group. If BP or HR is over 25-30 % baseline, an opioid or other pain medications will be used first, before increasing the dose of inhalational agent or propofol. If BP is low and PSI is on the low end, study team will lower the inhalational agent or propofol first. If the patient moves and BP and PSI are within the ranges, muscle relaxant may be given first unless the use of muscle relaxant is not allowed for the surgical reason. If both opioids and muscle relaxant adjustment fail to achieve the hemodynamic stability and immobility goal, then the study team will adjust the doses of inhalational agent or propofol.
* Time out performed

SEDATION The anesthesia provider will apply a Sedline Monitor to their forehead during the general anesthesia procedure. The anesthesia provider may use the data from the monitor to affect their anesthetic administration, or may cover the data from the monitor and only use conventional measures to guide anesthetic dosing in these control cases (blood pressure, heart rate, body movement, respiratory rate, MAC of inhalational agent), depending on what group into which the patient has been randomized.

* Start induction with Dex (3mcg/kg bolus of dexmedetomidine over 10 minutes, followed by a Dex infusion of 2mcg/kg/minute)
* Nasal cannula with ETCO2 placed
* Transport checklist (O2 tank full, Bag mask at head of bed, Airway bag, meds, transport monitor with battery, suction, emergency med bag) completed *only if MRI outside of Comer
* Patient transported to MRI
* Patient is placed on MRI table, monitors switched for MRI compatible monitors If additional medication is required for induction or movement artifact on MRI imaging, propofol bolus(es) or, in rare cases, fentanyl bolus(es), may be given as needed per standard sedation protocol. All sedation medications are documented in the medical record per protocol.

If BP or HR is over 25-30 % baseline, an opioid or other pain medications will be used first, before increasing the dose of inhalational agent or propofol. If BP is low and PSI is on the low end, study team will lower the inhalational agent or propofol first. If the patient moves and BP and PSI are within the ranges, muscle relaxant may be given first unless the use of muscle relaxant is not allowed for the surgical reason. If both opioids and muscle relaxant adjustment fail to achieve the hemodynamic stability and immobility goal, then the study team will adjust the doses of inhalational agent or propofol.

* MRI Scan completed
* Dex stopped and the time recorded. Dex infusion should continue until MRI completion, but weaning of Dex is allowed if deemed clinically appropriate. Weaning of Dex will be documented in the medical record as per sedation protocol.

RECOVERY

* After MRI is completed, patient is placed back on transport bed and monitors exchanged for transport monitors
* Patient transported back to sedation suite for recovery
* Sedline monitor is placed on patient.
* After 2-3 minutes of recording, patient receives study drug (caffeine citrate/placebo) at 10mL/kg over 5 minutes.
* Registered Nurse (RN) monitors patient per routine sedation protocol (every 5min vitals, Patient Sedation State Score [PSSS] score)
* Study team records time to awake
* Sedline monitor may be removed after patient is awake Once the general anesthesia procedure is over and the patient is recovering in PICU, the study team will meet with each patient and parent again, and use a standardized survey to ask about their satisfaction with their anesthetic, including questions about their post-operative pain and feelings of nausea or presence of vomiting. They should also be awake, be able to drink clear liquid, void and ambulate before discharge home with their parents.
* Study team records time to meet discharge criteria
* Patient discharged per routine protocol

FOLLOW-UP DAY 1 AFTER SEDATED MRI

* Patient receives call from sedation scheduler the next day per sedation team protocol
* Patient receives call from study team the next day via the standardized post-operative survey The study team will follow-up the next day with each patient's parent via phone call and ask the same survey questions to ensure resolution of their symptoms and timing of the resolution of their symptoms..

ELIGIBILITY:
Inclusion Criteria:

* Undergo Magnetic Resonance Imaging (MRI) scan
* Age ≥3 and ≤ 12 yr old
* Both Male and Female
* Weight ≤33.3 kg
* American Society of Anesthesiologists ASA) physical status 1-3
* No History of Arrhythmia (3-leads Electrocardiogram [EKG] applied before and after the sedation) or congenital heart disease
* Capable of obtaining consent from at least one parent
* No history of liver and kidney impairment
* No history of head trauma
* No prior history of difficulty with anesthesia
* No personal or family history of malignant hyperthermia

Exclusion Criteria:

* Age <3 or >12
* Weight >33.3 kg
* ASA physical status > 3
* History Arrhythmia, congenital heart disease, liver, and kidney diseases
* Prior difficulty with anesthesia
* Personal or family history of malignant hyperthermia
* Unable to obtain consent
* History of head trauma
* Female subjects who are pregnant

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Improve rate of wakefulness post surgery | Up to 2 hours
  Subject post-surgery wakefulness recovery with caffeine based on a modified Aldrete score

SECONDARY OUTCOMES:
Time needed to be able to return to tasks performance with purpose | Up to 2 hours
  Eyes open, normal response to verbal stimulation, crying/complaining, taking PO (if applicable)

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Xie, MD,PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xie Z, Fong R, Fox AP. Towards a potent and rapidly reversible Dexmedetomidine-based general anesthetic. PLoS One. 2023 Sep 26;18(9):e0291827. doi: 10.1371/journal.pone.0291827. eCollection 2023. PMID 37751454
- [Background] Xie Z, Fox AP. Rapid emergence from dexmedetomidine sedation in Sprague Dawley rats by repurposing an alpha2-adrenergic receptor competitive antagonist in combination with caffeine. BMC Anesthesiol. 2023 Feb 1;23(1):39. doi: 10.1186/s12871-023-01986-5. PMID 36721095
- [Background] Fong R, Wang L, Zacny JP, Khokhar S, Apfelbaum JL, Fox AP, Xie Z. Caffeine Accelerates Emergence from Isoflurane Anesthesia in Humans: A Randomized, Double-blind, Crossover Study. Anesthesiology. 2018 Nov;129(5):912-920. doi: 10.1097/ALN.0000000000002367. PMID 30044241
- [Background] Mason KP, Lerman J. Review article: Dexmedetomidine in children: current knowledge and future applications. Anesth Analg. 2011 Nov;113(5):1129-42. doi: 10.1213/ANE.0b013e31822b8629. Epub 2011 Aug 4. PMID 21821507